CLINICAL TRIAL: NCT06518603
Title: Randomized Controlled Trial of Caffeine Citrate in Preterm Infants at Risk of Apnea in Zambia
Brief Title: Caffeine Citrate in Preterm Infants at Risk of Apnea in Zambia
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University Teaching Hospital, Lusaka, Zambia (Other); Centre for Infectious Disease Research in Zambia (Other)
Responsible Party: Principal Investigator, Albert Manasyan, MD, MPH, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UAB-300013205; UAB Dixon End Chair/3102800 (Other: University of Alabama at Birmingham); 000533428-0004 (Other: INSIGHT)
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Premature Infant Disease; Apnea of Prematurity; Development, Infant
MeSH Terms: conditions — Apnea | interventions — caffeine citrate

STUDY DESIGN:
Intervention Model Description: Double blind, placebo-controlled, 1:1 parallel allocation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking will be maintained throughout the study and only the study pharmacists will be aware of the treatment group. The study pharmacist will prepare the 28-day supply of either caffeine citrate or placebo in indistinguishable clear solutions and same vials of equivalent volumes for the infant to continue at home. All other study staff, facility staff, follow-up staff, and family members will be masked to the treatment allocation. Identical vials will be prepared for the placebo arm with only a specific code written on the vials differentiating it from caffeine citrate. This code will be known only to the study pharmacist. Caffeine levels will not be checked routinely and checking levels will be discouraged to optimize masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Caffeine Citrate 20mg/kg/day (Experimental): Caffeine Citrate 20 mg/kg/day given orally once a day for 28 days. (2mg/ml)
  Interventions: Drug: Caffeine citrate 20mg/kg/day
- Placebo (Placebo Comparator): Sterile water 1ml/kg/day given orally once a day for 28 days.
  Interventions: Drug: Placebo-Sterile water 1ml/kg/day

INTERVENTIONS:
Drug: Caffeine citrate 20mg/kg/day — Caffeine citrate 20mg/kg/day given orally once daily for 28 days
  Arms: Oral Caffeine Citrate 20mg/kg/day
Drug: Placebo-Sterile water 1ml/kg/day — Placebo-sterile water 1mg/kg/day given orally once daily for 28 days
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if caffeine citrate prevents apneic events that result in sick visits in moderately preterm infants after discharge from the hospital. It will also learn if the use of caffeine leads to better developmental outcomes at 12 months of age.

Our research questions are:

1. Does continued treatment of moderately preterm newborns with caffeine citrate after hospital discharge prevent or decrease apneic events that result in sick visits?
2. Will the continued use of caffeine citrate lead to improved developmental outcomes among infants at 12 months of age?

Researchers will compare caffeine citrate to a placebo (a look-alike substance that contains no drug) to see if caffeine citrate prevents apneic spells which result in healthcare visits.

Parents of participants will:

1. Administer caffeine citrate 20mg/kg/day or a placebo (equivalent volume of sterile water) orally every day for up to 28 days after hospital discharge
2. Keep a diary of symptoms and any apneic events
3. Check in with researchers via telephone call once a week
4. Return to clinic for infant physical examination at 28 days
5. Return to the clinic for infant physical examination at 2 months

5. Return to clinic for infant neurodevelopmental examination with Ages and Stages Questionnaire at 12 months of age

DETAILED DESCRIPTION:
Once an infant has been deemed stable by the neonatologist and the neonatologist recommends discontinuing treatment for apnea of prematurity 5 days before hospital discharge as per standard of care, the parent/guardian will be approached for consent. Following consent, study participants will be randomized to either the Intervention Arm (20mg/kg/day caffeine citrate; 2mg/ml) dose and equal volume of placebo (sterile water) using trial-specific single dose caffeine/placebo vials. Upon the study participant's hospital discharge, the pharmacist will prepare the caffeine citrate and placebo relevant to the weight of the infant within 48 hours prior to discharge. The doses will not be adjusted for weight gain after discharge. Caffeine levels will not be checked routinely and checking levels will be discouraged to optimize masking.

While at the hospital, infants will receive the oral dose from government staff. Following hospital discharge, the parent/guardian will be given enough doses of caffeine or equivalent placebo for 28 days and will be asked to administer it to their infant orally daily, at the same time, until day 28. Unlike the intervention arm, all study participants randomized to the control arm (placebo) will discontinue receiving caffeine and will begin receiving placebo (sterile water) in the same volume orally as those in the intervention arm. The parent/guardian will also be given a booklet to register any apneic spells. The study RA will contact the parent/guardian on a weekly basis, up to day 28 and once at 2 months after hospital discharge for patient clinical monitoring and follow-up purposes.

Upon completion of the study at 12 months of life, all study participants will return to the hospital for neurodevelopmental screening using the Ages and Stages-3 Questionnaire for 12 months.

Data will be collected onto paper forms, which will then be entered into a REDCap Database, housed at the Centre for Infectious Disease Research in Zambia (CIDRZ) offices. Data forms will be kept in locked cabinets, retained and destroyed per incineration after 5 years. Access to the data forms and REDCap Database will be restricted to those with a need to know.

ELIGIBILITY:
Inclusion Criteria:

Newborns:

1. 29 0/7 to 33 6/7 weeks GA (or with a birth weight 1.0 to 2.0 kg if pregnancy dating is unreliable) admitted to the UTH NICU,
2. On methylxanthines with plans to discontinue on methylxanthine,
3. Off oxygen therapy for >48 hours at the time of evaluation for eligibility,
4. Receiving full daily feeds,
5. Deemed stable and ready to go off caffeine as recommended by the Neonatologist
6. 18+ years of age (parent)

Exclusion Criteria:

1. Newborns with neuromuscular conditions affecting respiration,
2. Major congenital malformations and genetic disorders,
3. Unable to obtain parental or guardian consent

Ages: 0 Days to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 340 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of apneic events | 28 days after discharge
  Documentation or report of apnea of prematurity [AoP], a condition exhibited by cessation of breathing for ≥20 or <20 seconds accompanied by bradycardia and/or cyanosis
Number of visits to healthcare professionals related to apneic events | 28 days after discharge
  Documentation or report of sick visit

SECONDARY OUTCOMES:
Number of all-cause sick visits | 2 months after discharge
  Documentation or report of sick visit
Percentage of neonatal mortality within 2 months after discharge | 2 months after discharge
  Documentation of neonatal death
Infant/Child Developmental Assessment | 12 months
  Score on "Ages and Stages Questionnaire" obtained at clinic visit

CONTACTS AND LOCATIONS:
Locations (1):
- University Teaching Hospital, Lusaka, Lusaka Province, Zambia